CLINICAL TRIAL: NCT02786381
Title: Idylla Respiratory (IFV-RSV) Panel Clinical Testing and Sample Collection Protocol in Support of 510(k) Premarket Submission
Brief Title: Idylla IFV-RSV Panel Clinical Testing
Acronym: RP1
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CODX0006NAP3001
Record Dates: First submitted 2015-12-04; First posted 2016-06-01 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-09

CONDITIONS: Respiratory Tract Infections; Influenza, Human; Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Nasal swabs (NS); Nasopharyngeal swabs (NP) in viral transport medium (VTM)
Oversight: Data Monitoring Committee: No

SUMMARY:
This clinical study will collect fresh samples and perform laboratory testing on fresh and archived samples as described in the protocol.

DETAILED DESCRIPTION:
The Idylla console, instrument, and Respiratory (IFV-RSV) Panel cartridge constitute the Idylla respiratory diagnostic system. The IFV-RSV Panel is an in vitro PCR-based molecular diagnostic assay for the simultaneous qualitative detection of nucleic acids for Influenza A (including H1, 2009 H1N1, H275Y mutation of 2009 H1N1, H3), Influenza B, and Respiratory Syncytial Virus (RSV) (A and B) on nasal swab (NS) direct to cartridge or nasopharyngeal swabs (NP) in viral transport media (VTM) in adults, adolescents, and children.

This clinical study will collect data in support of regulatory submission and the indications for use of the IFV-RSV panel and the Idylla diagnostic system. This protocol will demonstrate that the results of this assay, in conjunction with clinical information, may be used as an aid in the diagnosis of infection with Influenza A, Influenza B, and RSV in persons having both a high and low risk for respiratory viral infection.

During this study, participating sites will collect fresh samples, conduct a Reproducibility Study and test the fresh and previously collected frozen samples from individuals presenting with signs/symptoms of influenza like illness (ILI) and respiratory virus in accordance to the sample collection described in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* All Ages
* Subject, or legally authorized representative, has provided IRB/EC approved written Informed Consent, privacy (e.g. HIPAA) authorization when required and Assent where applicable prior to any study-related procedure(s) being performed
* Patient presenting with ILI and/or Signs/Symptoms of RSV Infection as defined in this protocol
* Onset of ILI and/or Signs/Symptoms of RSV Infection was ≤ 5 days prior to subject screening (Refer to the definitions for detailed descriptions of ILI and Signs/Symptoms of RSV infection)
* Clinician's determination that illness is due to a viral infection
* Subject agrees to allow study specimens to be used for future studies

Exclusion Criteria:

* Onset of Influenza Like Illness (ILI) and/or Signs/Symptoms of RSV Infection was > 5 days prior to subject screening (Refer the definitions for detailed descriptions of ILI and Signs/Symptoms of RSV infection)
* Subject received live intranasal attenuated influenza virus in last 3 weeks (e.g. FluMist, Fluenz)
* Subject received treatment with influenza directed antiviral (e.g. Zanamivir, oseltamivir (Tamiflu), amantadine, rimantadine) in the last 5 days
* The subject was previously enrolled in this study
* Clinician's determination that illness is NOT due to a viral infection (e.g. allergies)
* Subject had a nasal wash within last 8 hours. This exclusion includes any extraction of nasal secretions by nasal suctioning with fluid
* Subject does not agree to allow study specimens to be used for future research studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who present with ILI and/or signs/symptoms of RSV Infection who have met all the inclusion and none of the exclusion criteria are considered eligible to participate in the sample collection phase of this study. Specimens may be collected from subjects in either an inpatient or outpatient setting. An outpatient setting includes facilities such as emergency rooms associated with hospitals, large decentralized hospital/commercial labs, urgent cares and/or physician practices currently undertaking diagnostic testing. An inpatient setting is defined as a hospital where patients are admitted (does not include the emergency room associated with the hospital as this will be considered "outpatient" setting). Patient populations from the United States will be evaluated.
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Product performance as measured by positive and negative agreement to a predicate | Specimen collected during the IFV-RSV season 2015/2016 will be tested within 1 day of enrollment. The Product Performance will be assessed at study completion, an average of 6 months.
  Product Performance will be assessed based on samples collected in 2015/2016 season (average of 6 months) and archived samples.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Pattery, MD, Study Director — Janssen Diagnostics
Locations (1):
- Sacred Heart Hospital - Pensacola, Pensacola, Florida, United States